CLINICAL TRIAL: NCT01437566
Title: A Phase II, Double-Blind, Placebo Controlled, Randomized Study of GDC-0941 or GDC-0980 With Fulvestrant Versus Fulvestrant in Advanced or Metastatic Breast Cancer in Patients Resistant to Aromatase Inhibitor Therapy
Brief Title: Study of GDC-0941 or GDC-0980 With Fulvestrant Versus Fulvestrant in Advanced or Metastatic Breast Cancer in Participants Resistant to Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: GDC4950g; GO00769 (Other: Hoffmann-La Roche); 2010-023763-17 (EudraCT Number)
Record Dates: First submitted 2011-09-08; First posted 2011-09-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- GDC-0941 Matching Placebo + Fulvestrant (Arm E) (Placebo Comparator): Participants with PIK3CA mutation will receive fulvestrant 500 mg as 2 IM injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle and GDC-0941 matching placebo QD orally starting on Day 1 of Cycle 1, each cycle of 28 days. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Fulvestrant; Drug: GDC-0941 Matching Placebo
- GDC-0941-260 mg + Fulvestrant (Arm D) (Experimental): Participants with PIK3CA mutation will receive fulvestrant 500 mg as 2 IM injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle and GDC-0941 260 mg QD orally starting on Day 1 of Cycle 1, each cycle of 28 days. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Fulvestrant; Drug: GDC-0941
- GDC-0941-340 mg + Fulvestrant (Arm A) (Experimental): Participants will receive fulvestrant 500 milligrams (mg) as 2 intramuscular (IM) injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle and GDC-0941 340 mg once daily (QD) orally starting on Day 15 of Cycle 1, each cycle of 28 days. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Fulvestrant; Drug: GDC-0941
- GDC-0948 or GDC-0980 Matching Placebo + Fulvestrant (Arm C) (Placebo Comparator): Participants will be randomized in 1:1 ratio to receive GDC-0948 matching placebo or GDC-0980 matching placebo with fulvestrant. Participants will receive fulvestrant 500 mg as 2 IM injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle and GDC-0948 or GDC-0980 matching placebo QD orally starting on Day 15 of Cycle 1, each cycle of 28 days. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Fulvestrant; Drug: GDC-0941 Matching Placebo; Drug: GDC-0980 Matching Placebo
- GDC-0980-30 mg + Fulvestrant (Arm B) (Experimental): Participants will receive fulvestrant 500 mg as 2 IM injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle and GDC-0980 30 mg QD orally starting on Day 15 of Cycle 1, each cycle of 28 days. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Interventions: Drug: Fulvestrant; Drug: GDC-0980

INTERVENTIONS:
Drug: Fulvestrant — Participants will receive fulvestrant 500 mg as 2 IM injections of 250 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle, each cycle of 28 days until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
Drug: GDC-0941 — Participants will receive GDC-0941 260 mg (Part II) or 340 mg (Part I) QD orally from Day 1 or Day 15 of Cycle 1 until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Arms: GDC-0941-260 mg + Fulvestrant (Arm D); GDC-0941-340 mg + Fulvestrant (Arm A)
Drug: GDC-0941 Matching Placebo — Participants will receive GDC-0941 matching placebo QD orally from Day 1 or Day 15 of Cycle 1 until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Arms: GDC-0941 Matching Placebo + Fulvestrant (Arm E); GDC-0948 or GDC-0980 Matching Placebo + Fulvestrant (Arm C)
Drug: GDC-0980 — Participants will receive GDC-0980 30 mg (Part I) QD orally from Day 15 of Cycle 1 until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Arms: GDC-0980-30 mg + Fulvestrant (Arm B)
Drug: GDC-0980 Matching Placebo — Participants will receive GDC-0980 matching placebo QD orally from Day 15 of Cycle 1 until disease progression, intolerable toxicity, elective withdrawal from the study, study completion or termination.
  Arms: GDC-0948 or GDC-0980 Matching Placebo + Fulvestrant (Arm C)

SUMMARY:
This is a multicenter, international, randomized, double-blinded, placebo-controlled, Phase II trial. Participants with advanced breast cancer (ABC) or Metastatic Breast Cancer (MBC) who have experienced recurrence or progression of their disease while receiving aromatase inhibitor (AI) therapy or who have relapsed within 6 months after completing adjuvant AI therapy will be enrolled in Part I of this study. Participants with ABC or MBC who have received prior AI therapy and who have PIK3CA-mutant tumors will be enrolled in Part II of this study. Part I of the study will assess the effect of the addition of GDC-0941 to fulvestrant (Arm A) and of GDC-0980 to fulvestrant (Arm B) on progression free survival (PFS) compared with fulvestrant + placebo (Arm C). Part II of the study will examine the safety and tolerability and to estimate the effect of GDC-0941 in combination with fulvestrant (Arm D) on PFS versus fulvestrant + placebo (Arm E) in participants who received prior treatment with an AI and whose tumors contain a PIK3CA mutation.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* As per national or local treatment guidelines, endocrine therapy (i.e., fulvestrant) is recommended and treatment with cytotoxic chemotherapy is not necessary for participants, at time of entry into the study.
* Part I: Postmenopausal women with locally ABC or MBC whose disease relapsed during treatment with (or within 6 months after discontinuation of) an AI in the adjuvant setting or progressed during treatment with an AI in the metastatic setting.
* Part II: Postmenopausal women with locally ABC or MBC whose disease has progressed during or after treatment with an AI. Participants who discontinued the AI for toxicity rather than completion of regimen or for disease progression are not eligible
* Estrogen receptor (ER)-positive disease and human epidermal receptor 2 (HER2)-negative disease
* Participants must have measurable disease by response evaluation criteria in solid tumors (RECIST) version (v) 1.1 or bone-only disease with radiologic scans
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Prior treatment with fulvestrant, phosphoinositide 3-kinase (PI3K) inhibitor, or mechanistic target of rapamycin (mTOR) inhibitor for ABC or MBC
* Prior anti-cancer therapy or radiotherapy within 2 weeks prior to Day 1 of Cycle 1
* Prior treatment with greater than (>) one cytotoxic chemotherapy regimens or experienced recurrent or progressive disease on > two endocrine therapies for MBC
* Participants requiring anti-hyperglycemic therapy
* Clinically significant cardiac or pulmonary dysfunction
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant history of liver disease
* Active uncontrolled autoimmune disease or active inflammatory disease
* Immunocompromised status
* Need for current chronic corticosteroid therapy
* Pregnancy, lactation, or breastfeeding
* Current severe, uncontrolled systemic disease
* Symptomatic hypercalcemia
* Known untreated or active central nervous system (CNS) metastases
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or patients who have undergone potentially curative therapy with no evidence of disease and are deemed by the treating physician to be at low risk for recurrence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2011-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival as Assessed by the Investigator Per modified RECIST v 1.1 | From Screening to up to approximately 5 years (assessed at Screening, after 8, 16, 24 and 32 weeks of treatment, every 12 weeks thereafter until disease progression or initiation of other anti-cancer therapy)
Percentage of Participants with Adverse Events | Baseline to up to 30 days after the last dose of study drug (Approximately 5 years)

SECONDARY OUTCOMES:
Percentage of Participants with Objective Tumor Response (Complete Response [CR] or Partial Response [PR] as Assessed by the Investigator Per Modified RECIST v 1.1 | From Screening to up to approximately 5 years (assessed at Screening, after 8, 16, 24 and 32 weeks of treatment, every 12 weeks thereafter until disease progression or initiation of other anti-cancer therapy)
Percentage of Participants with Clinical Benefit Response Defined as PR, CR, or SD Per Modified RECIST v 1.1 | From Screening to up to approximately 5 years (assessed at Screening, after 8, 16, 24 and 32 weeks of treatment, every 12 weeks thereafter until disease progression or initiation of other anti-cancer therapy)
Duration of Confirmed Objective Response as Assessed by the investigator Per Modified RECIST v 1.1 | From Screening to up to approximately 5 years (assessed at Screening, after 8, 16, 24 and 32 weeks of treatment, every 12 weeks thereafter until disease progression or initiation of other anti-cancer therapy)
Percentage of Participants with PIK3CA Mutant Tumors | Baseline
Time to Maximum Plasma Concentration (Tmax) of GDC-0941 and GDC-0948 | Part 1:0-4 hour (hr) predose (PrD), 1,2,4 hr postdose (PoD) on Day 15 of Cycles 1 & 2, PrD on Cycle 1 Day 16, 0-4 hr PrD & 2 hr PoD on Cycle 6 Day 1; Part II:0-4 hr PrD, 2 hr PoD on Day 1 of Cycles 1 & 6, 0-4 hr PrD, 1, 2, 4 hr PoD on Cycle 2 Day 1
Maximum Plasma Concentration (Cmax) of GDC-0941 and GDC-0948 | Part 1:0-4 hr PrD, 1,2,4 hr PoD on Day 15 of Cycles 1 & 2, PrD on Cycle 1 Day 16, 0-4 hr PrD & 2 hr PoD on Cycle 6 Day 1; Part II:0-4 hr PrD, 2 hr PoD on Day 1 of Cycles 1 & 6, 0-4 hr PrD, 1, 2, 4 hr PoD on Cycle 2 Day 1
Area Under the Concentration Time Curve From Time Zero to 24 Hours Postdose (AUC0-24) of GDC-0941 and GDC-0948 | Part 1:0-4 hr PrD, 1,2,4 hr PoD on Day 15 of Cycles 1 & 2, PrD on Cycle 1 Day 16, 0-4 hr PrD & 2 hr PoD on Cycle 6 Day 1; Part II:0-4 hr PrD, 2 hr PoD on Day 1 of Cycles 1 & 6, 0-4 hr PrD, 1, 2, 4 hr PoD on Cycle 2 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Gallia Levy, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (115):
- United States (38):
  - Birmingham, Alabama
  - Hayward, California
  - Oakland, California
  - Roseville, California
  - Sacramento, California
  - San Francisco, California
  - San Jose, California
  - Santa Clara, California
  - South San Francisco, California
  - Vallejo, California
  - Walnut Creek, California
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Fort Myers, Florida
  - Jacksonville, Florida
  - St. Petersburg, Florida
  - Marietta, Georgia
  - Joliet, Illinois
  - Peoria, Illinois
  - Wichita, Kansas
  - Boston, Massachusetts
  - St Louis, Missouri
  - Basking Ridge, New Jersey
  - Hackensack, New Jersey
  - Commack, New York
  - New York, New York
  - Rockville Centre, New York
  - Sleepy Hollow, New York
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Tyler, Texas
  - Richmond, Virginia
- Argentina (2):
  - Buenos Aires
  - Santa Fe
- Australia (7):
  - Kogarah, New South Wales
  - Wahroonga, New South Wales
  - South Brisbane, Queensland
  - Bedford Park, South Australia
  - Woodville, South Australia
  - Frankston, Victoria
  - Parkville, Victoria
- Belgium (4):
  - Brussels
  - Edegem
  - Leuven
  - Liège
- Canada (3):
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan
- Chile (4):
  - Santiago
  - Temuco
  - Valparaíso
  - Viña del Mar
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Denmark (6):
  - Aarhus
  - Herlev
  - København Ø
  - Odense
  - Roskilde
  - Vejle
- Paris, France
- Germany (6):
  - Berlin
  - Düsseldorf
  - Freiburg im Breisgau
  - Hamburg
  - München
  - Trier
- Hong Kong (2):
  - Hong Kong
  - Pokfulam
- Israel (8):
  - Beersheba
  - Holon
  - Jerusalem
  - Kfar Saba
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Italy (7):
  - Napoli, Campania
  - Meldola, Emilia-Romagna
  - Milan, Lombardy
  - Monza, Lombardy
  - Pisa, Tuscany
  - Prato, Tuscany
  - Terni, Umbria
- Malaysia (3):
  - George Town
  - Kuala Lumpur
  - Tanjung Bungah
- León, Mexico
- New Zealand (3):
  - Christchurch
  - Hamilton
  - Wellington
- Lima, Peru
- Russia (4):
  - Chelyabinsk
  - Kazan'
  - Moscow
  - Voronezh
- Singapore, Singapore
- Seoul, South Korea
- Spain (4):
  - Barcelona, Barcelona
  - Lleida, Lerida
  - Valencia, Valencia
  - Zaragoza, Zaragoza
- Thailand (2):
  - Patumwan
  - Songkhla
- United Kingdom (4):
  - Brighton
  - Cardiff
  - London
  - Stoke-on-Trent

REFERENCES:
- [Derived] Krop IE, Mayer IA, Ganju V, Dickler M, Johnston S, Morales S, Yardley DA, Melichar B, Forero-Torres A, Lee SC, de Boer R, Petrakova K, Vallentin S, Perez EA, Piccart M, Ellis M, Winer E, Gendreau S, Derynck M, Lackner M, Levy G, Qiu J, He J, Schmid P. Pictilisib for oestrogen receptor-positive, aromatase inhibitor-resistant, advanced or metastatic breast cancer (FERGI): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2016 Jun;17(6):811-821. doi: 10.1016/S1470-2045(16)00106-6. Epub 2016 May 4. PMID 27155741